CLINICAL TRIAL: NCT07007910
Title: A Phase I Clinical Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of HSK46575 Tablets in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Phase I Study of HSK46575 in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK46575-101
Record Dates: First submitted 2025-05-22; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: m CRPC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase Ia (Dose Escalation Part): HSK46575 (Experimental): Phase 1a (Dose Escalation Part): dose escalation of HSK46575 at various dose levels
  Interventions: Drug: HSK46575
- Phase Ia (Extension Part): HSK46575 (Experimental): Phase 1a (Part B): dose extention of HSK46575 at certain dose levels
  Interventions: Drug: HSK46575
- Phase Ib: HSK46575 (Experimental): Phase 1b: dose expansion for HSK46575 at dose of RP2D（Recommended Phase II Dose）
  Interventions: Drug: HSK46575

INTERVENTIONS:
Drug: HSK46575 — co-administered with glucocorticoid and fludrocortisone, orally daily

SUMMARY:
This is a phase I, open-label, dose-escalation and expansion study to evaluate the safety, tolerability, PK（pharmacokinetics） and PD（pharmacodynamics） of HSK46575 when given orally in patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
The study will contain two phases: Phase Ia is dose escalation phase and Phase Ib is dose expansion phase.

Phase Ia will contain two part: Dose Escalation Part and Extension Part. Dose Escalation Part based on the "3+3" design for dose escalation and safety evaluation requirements. Patient cohorts at selected doses may be extended to further investigate the tolerability, PK and PD of HSK46575. The number of patients to be enrolled will be up to 10 subjects in each Extension Part cohort. Approximately 30 subjects will be enrolled in Phase Ia.

Phase Ib no less than 60 subjects will be enrolled in each expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged ≥18 years;
2. ECOG (Eastern Cooperative Oncology Group) 0-1, expected survival of ≥ 3 months;
3. Histology or cytology confirmed adenocarcinoma of the prostate;
4. Radiological evidence of metastatic bone or soft tissue lesions;
5. Ongoing medical castration or previous surgical castration;
6. Testosterone at castration level during screening;
7. Prior to screening, subjects with evidence of disease progression while receiving ADT (androgen deprivation therapy);
8. Had progressed on at least one novel endocrine therapy, and had progressed on at least one taxane-based chemotherapy (or those who are intolerant or refuse chemotherapy);
9. The functional level of organs must meet the requirements.

Exclusion Criteria:

1. Subjects with known hypersensitivity to the active ingredient or excipients of HSK46575 Tablets;
2. Subjects who have received any antitumor therapy within 4 weeks (or 5 half-lives, whichever is shorter) prior to the first dose; or treatment with nitrosoureas, bicalutamide, or nilutamide within 6 weeks (or 5 half-lives, whichever is shorter) prior to the first dose;
3. Subjects whose toxicity from prior anticancer therapy remains > Grade 1 before the first dose;
4. Subjects who have used strong or moderate CYP3A4 inhibitors or inducers, CYP2C9 sensitive substrates, and OCT2 or MATE1 substrates within 14 days or 5 half-lives prior to the first dose of the investigational drug, whichever is longer;
5. Subjects who have undergone Grade 3-4 surgery;
6. Subjects who plan to receive any other antitumor therapy during the study ;
7. Subjects with active metastases to central nervous system;
8. Subjects with serious bone damage caused by prostate cancer bone metastasis as assessed by the investigators;
9. Within 6 months before the first dose, subjects had concurrent pituitary or adrenal dysfunction;
10. Subjects with uncontrolled hypertension;
11. Subjects with central nervous system disorders such as epilepsy and multiple sclerosis;
12. Subjects with active cardiac disease within 6 months prior to the first dose, or a history of arterial or venous thromboembolism;
13. Subjects with a QTc interval prolongation to >470 ms during the screening period calculated by the Fridericia formula；
14. Subjects with a history of other malignancies;
15. Subjects with a history of immunodeficiency;
16. Subjects with active HBV, HCV, or syphilis infection;
17. Subjects who have participated in other clinical studies within 4 weeks before the first dose;
18. Other conditions.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Within first 28 days of treatment
  Highest dose level at which under 33% of patients in a cohort experience DLT（dose limiting toxicity）

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No